CLINICAL TRIAL: NCT06234865
Title: The Effect of Technology-based Constipation Prevention Training on Constipation Management in Hospitalised Orthopaedic Patients
Brief Title: Technology-based Constipation Prevention Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Sinan Aydoğan, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MehmetAkifU-SBF-SA-1
Record Dates: First submitted 2024-01-15; First posted 2024-01-31 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Constipation
Keywords: constipation; nursing; orthopedic
MeSH Terms: conditions — Constipation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in the control group will receive the routine care of the orthopaedic clinic and education with a brochure about preventing constipation.
  Interventions: Other: Control Group
- Video Education Group (Experimental): Patient in the experimental group will receive the routine care of the orthopaedic clinic and a video education about preventing constipation.
  Interventions: Other: Video Education Group

INTERVENTIONS:
Other: Control Group — Patients in the control group will receive standard education plus a brochure education. Standard education includes education provided by the doctor, nurse and/or physiotherapist before and after surgery. The brochure education includes information about constipation and interventions that can be used to prevent constipation such as nutrition, fluid intake, physical activity, leg exercises, abdominal massage, and toilet habits.
  Arms: Control Group
Other: Video Education Group — Patients in the experimental group will receive standard education plus a video education. Standard education includes education provided by the doctor, nurse and/or physiotherapist before and after surgery. The video education includes information about constipation and interventions that can be used to prevent constipation such as nutrition, fluid intake, physical activity, leg exercises, abdominal massage, and toilet habits.
  Arms: Video Education Group

SUMMARY:
The aim of this study is to determine the effect of technology-assisted constipation prevention training on the management of constipation in hospitalised orthopaedic patients. This is a quasi-experimental study. The population of the study will consist of patients admitted to the Orthopaedic Clinic of Burdur State Hospital between January 2024 and November 2024. The sample of the study is planned to consist of patients over 18 years of age, who are able to communicate, who do not have sensory loss related to advanced vision and hearing, who do not have psychiatric disorders at a level that prevents communication, and who are hospitalised at the Orthopaedic Clinic and who volunteer to participate in the research. Data for the study will be collected using the "Patient Introduction Form", "Constipation Risk Assessment Scale (CRAS)", "Bristol Stool Consistency Scale", "Use of Constipation Prevention Methods Form", "Constipation Education Questionnaire", "Constipation Severity Scale". During the implementation of the research, it is planned to form two groups, the first 35 patients in the control group and the second 35 patients in the experimental group, from the patients hospitalised in the Orthopaedic Clinic. The data will be collected at 3 times: (1) before the training, (2) 2 weeks after the training, (3) 4 weeks after the training. The data will be digitalised in the SPSS 23 package and the necessary statistical analyses will be performed.

DETAILED DESCRIPTION:
Objective: The aim of this study is to determine the effect of technology-assisted constipation prevention training on constipation management for patients admitted to an orthopaedic clinic.

Method This is a quasi-experimental study. The population of the study will consist of patients admitted to the Orthopaedic Clinic of Burdur State Hospital between January 2024 and November 2024. The sample of the study will consist of patients over the age of 18, who are able to communicate, who do not have advanced sensory loss related to vision and hearing, who do not have psychiatric disorders at a level that prevents communication, and who are admitted to the Orthopaedic Clinic and volunteer to participate in the study.

The study population consisted of patients admitted to the orthopaedic service. To calculate the sample size, an α error of 0.05 and a power of 0.95 were set using G power 3.1 software, based on previous studies with a similar design. As a result, a total of 70 patients were needed for this study after accounting for a 10% drop-out rate.

Data collection The data of the study will be collected by "Patient Introduction Form", "Constipation Risk Assessment Scale (CRAS)", "Bristol Stool Consistency Scale", "Use of Constipation Prevention Methods Form", "Constipation Education Questionnaire", "Constipation Severity Scale".

The "Patient Introduction Form", "Use of Constipation Prevention Methods Form" and "Constipation Education Questionnaire" will be prepared by the researchers according to the information in the literature.

Implementation of the research During the implementation of the research, it is planned to form two groups, the first 35 patients in the control group and the second 35 patients in the experimental group, from the patients admitted to the Orthopaedic Clinic.

The 'Patient Introduction Form', 'Constipation Risk Assessment Scale (CRAS)', 'Bristol Stool Consistency Scale' and 'Constipation Severity Scale' will be used for the patients in the control group. The Bristol Stool Consistency Scale will be given to patients to facilitate telephone follow-up. Patients' constipation management will be assessed twice, two weeks and one month after the interview day. The Bristol Stool Consistency Scale, the Use of Constipation Prevention Methods Form and the Constipation Severity Scale will be completed. A constipation prevention booklet is given by the nurses as part of routine clinic care.

The ''Patient Introduction Form'', ''Constipation Risk Assessment Scale (CRAS)'', ''Bristol Stool Consistency Scale'' and ''Constipation Severity Scale'' will be applied to the patients in the experimental group. Unlike the control group, the patient will be asked to watch an educational video about constipation using a tablet. In addition, the patient will be given a constipation education booklet. A 'Constipation Education Question Form' will be completed after the training. The Bristol Stool Consistency Scale will be given to patients to facilitate telephone follow-up. As in the control group, the patients' constipation management will be evaluated twice, two weeks and one month after the day of the patient interview. The Bristol Stool Consistency Scale, the Visual Comparison Scale, the Use of Constipation Prevention Methods Form and the Constipation Severity Scale will be completed. Routine care is provided by nurses in the clinic.

Analyzing the Data The data will be digitalised in the SPSS 23 package and the necessary statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years of age
* be hospitalised at the Orthopaedic Clinic
* to be able to read and write
* be willing to participate in the research
* having a moderate or high risk of constipation according to the Constipation Risk Assessment Scale (CRAS) or being constipated

Exclusion Criteria:

* has bowel obstruction, irritable bowel syndrome, inflammatory bowel disease, hernia and bowel cancer
* has a psychiatric disorder at a level that prevents communication
* Difficulty in understanding and speaking Turkish
* Severe sensory loss related to vision and hearing
* Having a colostomy or ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Bristol Stool Consistency Scale | 1 month
  The Bristol Stool Consistency Scale was developed by Lewis and Heaton (1997) at the University of Bristol in the United Kingdom and is based on the visualisation of seven stool shapes to determine stool consistency. According to the Bristol Stool Consistency Scale, type 1 and type 2 indicate constipation, type 3 and type 4 indicate normal stools, and type 5, type 6 and type 7 indicate diarrhoea. It is recognised that there is a direct relationship between the shape of the stool and the length of time it remains in the colon. The form has been designed to enable patients to visually identify the consistency of stool at each defecation. It can be used with illiterate patients. The form is completed by the researcher face-to-face with the patient during the application process.
Costipation Severity Scale | 1 month
  The Turkish validity and reliability of the CSS, which was developed by Varma et al. in 2008, was conducted by Kaya and Turan (2010).The CSS is a scale to determine the frequency, intensity, and difficulty of defecation. This scale was also designed to measure constipation symptoms. The scale consists of 16 questions. The CSS has three sub-dimensions: Bowel Obstruction, Colon Laziness and Pain. The score that can be obtained from the Faecal Obstruction sub-dimension is 0-28, the score that can be obtained from the Constipation sub-dimension is 0-29, and the score that can be obtained from the Pain sub-dimension is 0-16. The lowest total score that can be obtained from the CSS is 0 and the highest score is 73. The high score obtained from the scale indicates that the symptoms are severe.

SECONDARY OUTCOMES:
Constipation Education Questionnaire | 1 month
  This form, developed by the researchers, contains a total of 5 questions to measure the patient's level of understanding and satisfaction with the education provided.
Use of constipation prevention methods | 1 month
  This investigator-developed form included 6 questions about the patients' diet, fluid intake, whether they used abdominal massage, leg exercises, physical activity, and whether they delayed bowel movements.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Aydoğan, Ph.D., Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur State Hospital, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kutlu AK, Yilmaz E, Cecen D, Eser E. The reliability and validity of the Turkish version of the constipation risk assessment scale. Gastroenterol Nurs. 2011 May-Jun;34(3):200-8. doi: 10.1097/SGA.0b013e31821ab553. PMID 21637085
- [Background] Kaya, N. ve Turan, N. (2011). Konstipasyon Ciddiyet Ölçeğinin güvenilirlik ve geçerliliği. Türkiye Klinikleri Journal of Medical Sciences, 31(6), 1491- 1501. doi: 10.5336/medsci.2010-22198
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672